CLINICAL TRIAL: NCT06598644
Title: Comparison of Cervical Sustained Natural Apophyseal Glide and Instrument Assisted Soft Tissue Mobilization on Mechanical Neck Pain
Brief Title: Comparison of Sustained Natural Apophyseal Glide &Amp; Instrument Assisted Soft Tissue Mobilization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01933 Maha Mustafa
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Mechanical Neck Pain
Keywords: cervical SNAGS; Instrument assisted soft tissue mobilization; ergon technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical SNAGS (C3-C7) + Conventional PT (Other)
  Interventions: Other: Cervical SNAGS (C3-C7) + Conventional PT
- IASTM (ergon) + Conventional PT (Active Comparator)
  Interventions: Other: IASTM (ergon) + Conventional PT

INTERVENTIONS:
Other: Cervical SNAGS (C3-C7) + Conventional PT — Cervical SNAGS at C3-C7 with active movements of lateral flexion and rotation with overpressure at the end range. .Frequency: 10 reps 3 times/week for 3 consecutive weeks Intensity: starting from 20% to 50% resistance across barrier provided by Physical therapist Conventional PT including 1-hot pack for 10 minutes 2-Cervical Stretchings for levator scapulae and sternocleidomastoid 3-cervical isometric exercises, 4. Cervical Range of motion exercises
  Arms: Cervical SNAGS (C3-C7) + Conventional PT
Other: IASTM (ergon) + Conventional PT — IASTM, ergon applied at levator scapulae and sternocleidomastoid muscle, with 30 strokes at an angle. After that icing done at the levator scapulae and sternocleidomastoid muscle for 5-10 minutes using cold pack.
  Arms: IASTM (ergon) + Conventional PT

SUMMARY:
The aim of this randomized controlled trial is to evaluate and compare the effectiveness of two therapeutic techniques-Cervical Sustained Natural Apophyseal Glide (SNAG) and Instrument-Assisted Soft Tissue Mobilization (IASTM)-in the treatment of mechanical neck pain. The trial seeks to determine which method is more effective in reducing pain, improving range of motion, and enhancing overall neck function in individuals suffering from mechanical neck pain.

DETAILED DESCRIPTION:
: Mechanical neck pain refers to pain that originates from the structures of the neck, including muscles, ligaments, joints, or intervertebral discs. Mechanical neck pain has a lifetime prevalence of about 30% to 50% in the general adult population. At any given point in time, the prevalence of neck pain is estimated to be between 10% and 20%. It is often characterized by pain that worsens with specific neck movements or sustained postures and can be associated with muscle tightness, stiffness, or reduced range of motion. Although various muscles and joints around the cervical region can be affected but sternocleidomastoid and levator scapulae are one the commonly affected muscles, with lower cervical spine (C3-C7) being affected.

.Cervical SNAGs are a manual therapy technique that involves the application of sustained glides to the cervical spine while the patient performs specific movements. This technique is designed to address joint dysfunction, improve range of motion, and reduce pain .IASTM involves the use of specialized tools to apply controlled micro trauma to soft tissues, such as muscles, fascia, and tendons. This technique is used to address soft tissue dysfunction and improve tissue quality.

IASTM helps to break down scar tissue and adhesions that can form after injury or due to chronic poor posture, leading to improved tissue mobility and function. The controlled micro trauma induced by IASTM stimulates a localized inflammatory response, which promotes tissue repair and remodeling The technique enhances local blood circulation, bringing nutrients and oxygen to the affected area and aiding in the removal of metabolic waste products. The technique can modulate pain through mechanical stimulation of sensory receptors in the soft tissues, leading to pain relief. By addressing soft tissue restrictions, IASTM can help restore normal range of motion in the cervical spine. IASTM can be performed 2-3 times per week, depending on the severity of symptoms and patient response. Proper application of IASTM can help reduce muscle tension, improve range of motion, and alleviate pain in the levator scapulae and sternocleidomastoid muscles. Aftercare instructions, include hydration and avoiding immediate strenuous activity. The rationale for the use of Cervical SNAGs is to help to mobilize the facet joints of the cervical spine, which can become stiff due to poor posture, injury, or degenerative changes. he technique can alleviate pain by reducing joint stiffness and improving the alignment of the cervical vertebrae. By improving joint mobility, SNAGs can help normalize muscle function and reduce muscle spasms or tension. Patients perform active movements during SNAGs, which helps integrate the improved joint mobility into functional activities, leading to better outcomes in daily tasks. The technique enhances proprioceptive feedback from the cervical spine, helping patients achieve better neck posture and movement control. The rationale for the use of IASTM lies in breaking down scar tissue and adhesions, promoting tissue healing and remodeling, improving range of motion, reducing pain, enhancing blood flow and circulation, improving proprioception and neuromuscular control, non-Invasive and complementary approach.

ELIGIBILITY:
Inclusion Criteria:

* • Both genders (males and females)

  * Age between 20 and 45 years
  * History of neck pain >3 month, with tenderness on palpation present on sternocleidomastoid and Levator scapulae muscles and pain aggravated by activities involving turning head towards the side
  * Patients with pain on NPRS (at least 3)

Exclusion Criteria:

* • patients with recent injuries or surgeries in and around the neck region

  * Cervical nerve root lesion (radiculopathy)
  * Traumatic injuries like whiplash injury
  * malignancy in and around the neck region
  * rheumatoid arthritis
  * pregnant females
  * cervicogenic headache
  * Patients with unwillingness or inability to provide informed consent
  * Current participation in another neck pain treatment program

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Neck disability index (NDI) | 3 weeks
  The NDI is a Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
Numeric Pain Rating Scale NPRS | 3 weeks
  The NPRS is a segmented numeric version of the visual analog scale which is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Universal goniometer | 3 weeks
  It is an instrument that measures the range of motion at a joint.

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No